CLINICAL TRIAL: NCT02440035
Title: Phase 1, First in Human Study to Evaluate the Safety, Tolerability and Immunogenicity of Ad35.RSV.FA2 Regimens Boosted With Ad26.RSV.FA2 in Healthy Adult Volunteers
Brief Title: A Study to Evaluate the Safety, Tolerability and Immunogenicity of Ad35.RSV.FA2 Regimens Boosted With Ad26.RSV.FA2 in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Crucell Holland BV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CR107409; VAC18192RSV1001 (Other: Crucell Holland BV)
Record Dates: First submitted 2015-05-07; First posted 2015-05-12 (Estimated); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Healthy Participants
Keywords: Healthy Participants; Ad35.RSV.FA2; JNJ-61187191

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

ARMS (4):
- Group 1 (Experimental): Two subsequent Intramuscular injections of Ad35.RSV.FA2 (1x10^11 virus particles [vp]) on Day 1, Day 85 and an intramuscular injection of Ad26.RSV.FA2 (5x10^10 vp) on Day 169.
  Interventions: Biological: Ad35.RSV.FA2; Biological: Ad26.RSV.FA2
- Group 2 (Experimental): Intramuscular injection of Ad35.RSV.FA2 (1x10^11 vp) on Day 1, an intramuscular injection of placebo control on Day 85 and an injection of Ad35.RSV.FA2 (1x10^11 vp) on Day 169.
  Interventions: Biological: Ad35.RSV.FA2; Drug: Placebo
- Group 3 (Experimental): One intramuscular injection of Ad35.RSV.FA2 (1x10^11 vp) on Day 1 and an intramuscular injection of placebo control on Day 85 and an intramuscular injection of Ad26.RSV.FA2 (5x10^10 vp) on Day 169.
  Interventions: Biological: Ad35.RSV.FA2; Biological: Ad26.RSV.FA2; Drug: Placebo
- Group 4 (Experimental): Two subsequent intramuscular injections of placebo control on Day 1, Day 85 and an intramuscular injection of Ad26.RSV.FA2 (5x10^10 virus particles [vp]) on Day 169.
  Interventions: Biological: Ad26.RSV.FA2; Drug: Placebo

INTERVENTIONS:
Biological: Ad35.RSV.FA2 — Participants will receive Intramuscular injection of Ad35.RSV.FA2 (1x10^11) virus particles on Day 1 and 85 in Group 1. Intramuscular injection of Ad35.RSV.FA2 (1x10^11) virus particles on Day 1 and 169 in Group 2. Intramuscular injection of Ad35.RSV.FA2 (1x10^11) virus particles on Day 1 in Group 3.
  Other Names: JNJ-61187191-AAA
  Arms: Group 1; Group 2; Group 3
Biological: Ad26.RSV.FA2 — Participants will receive Intramuscular injection of Ad26.RSV.FA2 (5x10^10 virus particles [vp]) on Day 169 in Group 1. Intramuscular injection of Ad26.RSV.FA2 (5x10^10) virus particles on Day 169 in Group 3. Intramuscular injection of Ad26.RSV.FA2 (5x10^10) virus particles on Day 169 in Group 4.
  Other Names: JNJ-61187165-AAA
  Arms: Group 1; Group 3; Group 4
Drug: Placebo — Participants will receive intramuscular injection of placebo (sterile formulation buffer) on Day 85 in Group 2. One intramuscular injections of placebo on Day 85 in Group 3. Two intramuscular injections of placebo on Day 1, and Day 85 in Group 4.
  Arms: Group 2; Group 3; Group 4

SUMMARY:
The purpose of this study is to assess the safety and tolerability of intramuscular homologous and heterologous prime-boost regimens of Ad35.RSV.FA2 (human adenovirus-vectored vaccine candidate) and Ad26.RSV.FA2 in healthy participants.

DETAILED DESCRIPTION:
This is a single-center, randomized (study medication assigned to participants by chance), placebo-controlled (an inactive substance; a pretend treatment [with no drug in it] that is compared in a clinical trial with a drug to test if the drug has a real effect), double-blind (neither the researchers nor the participants know what treatment the participant is receiving) and Phase 1 study in healthy participants. The study comprises a 4-week screening period; vaccination for each participant on Days 1, 85, and, 169; a 28-day follow-up period performed after each vaccination and a final visit at Day 323 or 351. Participants will be randomly assigned to one of the 4 treatment groups (Group 1/2/3/4) to receive either Ad35.RSV.FA2 or Ad26.RSV.FA2 or placebo. The study duration will be approximately 52 weeks. Blood samples for immunogenicity will be collected. Participant's safety will be evaluated throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be in good health, without significant medical illness, on the basis of physical examination, medical history, vital signs measurement, and 12-lead electrocardiogram (ECG) performed at screening
* Participant must meet protocol defined laboratory criteria within 28 days before Day 1
* Before randomization, a woman must be either; Not of childbearing potential: postmenopausal or surgically sterilized; of childbearing potential and practicing an effective method of birth control before vaccination and through 3 months after the last vaccination. Women, who are not heterosexually active at screening, must agree to utilize highly-effective methods of birth control if they become heterosexually active until 3 months after receiving the last dose of study vaccine
* A woman must have a negative serum pregnancy test (beta-human chorionic gonadotropin [beta-hCG]) at the screening visit, and a negative urine pregnancy test pre-vaccination on Day 1
* A woman must agree not to donate eggs (ova, oocytes) for the purposes of assisted reproduction until 3 months after receiving the last dose of study vaccine. A man must agree not to donate sperm until 3 months after receiving the last dose of study vaccine

Exclusion Criteria:

* Participant has a body mass index (BMI) less than or equal to (<=)19 and greater than or equal to (>=30) kilogram per square meter (kg/m2)
* Participant has any clinically significant acute or chronic medical condition that, in the opinion of the investigator, would preclude participation (e.g. history of seizure disorders, bleeding/clotting disorder, autoimmune disease, active malignancy, poorly controlled asthma, active tuberculosis or other systemic infections)
* Participant has had major surgery within the 4 weeks prior to randomization or has planned major surgery through the course of the study
* Participant has chronic active hepatitis B or hepatitis C infection, documented by hepatitis B surface antigen and hepatitis C antibody, respectively
* Participant has human immunodeficiency virus (HIV) type 1 or type 2 infection

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2015-04-21 (Actual); Primary Completion 2016-06-09 (Actual); Study Completion 2016-06-09 (Actual)

PRIMARY OUTCOMES:
Solicited Local and Systemic Adverse Events (AEs) | Up to 8 days after each vaccination
  Solicited AEs are precisely defined events that participants are specifically asked about and which are noted by participants through the participant diary.
Unsolicited AEs | From Signing of informed consent up to 28 days after each vaccination
  Unsolicited AEs will be reported by the participant from when the informed consent form (ICF) is signed until 28 days after each vaccination, or early discontinuation.
Serious Adverse Events (SAEs) | Up to Day 337
  A serious adverse event (SAE) is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly

SECONDARY OUTCOMES:
Determination of Respiratory Syncytial Virus (RSV)-Specific Humoral Immune Response | Day 1 (predose) up to day 337
  Determine induction and persistence of humoral immune response against RSV F-protein.
To Assess RSV-specific Cellular Immune Response | Day 1 (predose) up to day 337
  Assess the quantity and quality of the elicited cellular immune response.

CONTACTS AND LOCATIONS:
Overall Officials: Crucell Holland BV Clinical Trial, Study Director — Crucell Holland BV
Locations (1):
- Miami, Florida, United States